CLINICAL TRIAL: NCT05104255
Title: Factors Influencing the Neonatal Outcomes in Twin Pregnancies Undergoing Cesarean Section: a Cross-sectional Study
Brief Title: Neonatal Outcomes in Twin Pregnancies
Status: Completed | Type: Observational
Sponsor: Derince Training and Research Hospital (Other)
Collaborators: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Hande Gurbuz, Medical Doctor, Associate Professor, Principal Investigator, Bursa Yuksek Ihtisas Training and Research Hospital
Other Study IDs: 2019/05-26
Record Dates: First submitted 2021-10-21; First posted 2021-11-02 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Twin Pregnancy; Neonate
Keywords: General anesthesia; Neonate; Obstetric anesthesia; Pregnancy Outcomes; Spinal anesthesia; Twins; Twin pregnancy
MeSH Terms: interventions — Anesthesia, Spinal; Anesthesia, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Twin neonates: The demographic data and characteristics of the twins were evaluated.
  Interventions: Procedure: Spinal anesthesia; Procedure: General anesthesia

INTERVENTIONS:
Procedure: Spinal anesthesia — Twins delivered under under spinal anesthesia
Procedure: General anesthesia — Twins delivered under general anesthesia

SUMMARY:
Multiple pregnancies are associated with increased maternal and fetal risks compared to singleton pregnancies. Additionally, the cesarean section rate is quite high in multiple pregnancies. This study aimed to evaluate maternal and fetal characteristics and factors affecting fetal outcomes in twin pregnancies delivered by cesarean section.

DETAILED DESCRIPTION:
While the frequency of multiple pregnancies varies significantly among societies and individuals, especially in middle and high-income countries, the rate of multiple pregnancies has shown a significant rise worldwide in recent years, with the frequent use of assisted reproductive techniques, which has increased due to an increase in maternal age and a decrease in fertility. As a result, multiple pregnancies constitute approximately 2-4% of all births.

Multiple pregnancies are known to be associated with increased maternal and fetal risks compared to singleton pregnancies. While maternal mortality associated with a twin pregnancy is 2.5 times higher than in singleton pregnancy, adverse neonatal outcomes such as perinatal mortality, fetal growth restriction, and low birth weight are two to three times higher in twins than in singleton newborns. Moreover, neonatal near-miss, which refers to cases that almost resulted in death, is associated with multiple pregnancies.

For all these reasons, the planned cesarean section has been advocated over planned vaginal delivery to reduce the risk of adverse neonatal outcomes (especially for the second-born twin). However, cesarean delivery is known to be associated with a higher risk of maternal morbidity and poor neonatal outcomes. The vast majority of these risks are related to maternal hypotension, prolonged uterine-incision-to-delivery time, and general anesthesia. From this perspective, we aimed to evaluate maternal and fetal characteristics and factors affecting fetal outcomes in twin pregnancies delivered by cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Twin pregnancies
* Parturients delivered by cesarean section

Exclusion Criteria:

* The triplets or more multiple pregnancies
* Twins delivered through the vaginal route were excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The twin newborns were delivered by cesarean section.
Sampling Method: Non-Probability Sample
Enrollment: 527 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Appearance-Pulse-Grimace-Activity-Respiration-1st minute (worst:0; best:10) | 1 minute
  Appearance-Pulse-Grimace-Activity-Respiration (APGAR) score at the 1st minute after delivery
Appearance-Pulse-Grimace-Activity-Respiration-5th minute (worst:0; best:10) | 5 minute
  Appearance-Pulse-Grimace-Activity-Respiration (APGAR) score at the 5th minute after delivery
The Number of Participants Admitted to Neonatal Intensive Care Unit | 1 hour
  Admission to Neonatal Intensive Care Unit after delivery
The Number of Participants needed for Mechanical ventilation | 28 days
  The need for non-invasive and invasive mechanical ventilation
The Rate of Death | 28 days
  Neonatal mortality within the first 28 days after birth.

CONTACTS AND LOCATIONS:
Overall Officials: Hande Gurbuz, Assoc. Prof., Study Director — Bursa Yuksek Ihtisas Training and Research Hospital

IPD SHARING:
Plan to Share IPD: Yes
Individual, de-identified participant data will be shared with the researchers who provide a methodologically sound proposal.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning nine months following a possible publication and ending after one year.

REFERENCES:
- [Result] Young BC, Wylie BJ. Effects of twin gestation on maternal morbidity. Semin Perinatol. 2012 Jun;36(3):162-8. doi: 10.1053/j.semperi.2012.02.007. PMID 22713496
- [Result] Santana DS, Surita FG, Cecatti JG. Multiple Pregnancy: Epidemiology and Association with Maternal and Perinatal Morbidity. Rev Bras Ginecol Obstet. 2018 Sep;40(9):554-562. doi: 10.1055/s-0038-1668117. Epub 2018 Sep 19. PMID 30231294
- [Result] Cheong-See F, Schuit E, Arroyo-Manzano D, Khalil A, Barrett J, Joseph KS, Asztalos E, Hack K, Lewi L, Lim A, Liem S, Norman JE, Morrison J, Combs CA, Garite TJ, Maurel K, Serra V, Perales A, Rode L, Worda K, Nassar A, Aboulghar M, Rouse D, Thom E, Breathnach F, Nakayama S, Russo FM, Robinson JN, Dodd JM, Newman RB, Bhattacharya S, Tang S, Mol BW, Zamora J, Thilaganathan B, Thangaratinam S; Global Obstetrics Network (GONet) Collaboration. Prospective risk of stillbirth and neonatal complications in twin pregnancies: systematic review and meta-analysis. BMJ. 2016 Sep 6;354:i4353. doi: 10.1136/bmj.i4353. PMID 27599496
- [Result] National Collaborating Centre for Women's and Children's Health (UK). Multiple Pregnancy: The Management of Twin and Triplet Pregnancies in the Antenatal Period. London: RCOG Press; 2011 Sep. Available from http://www.ncbi.nlm.nih.gov/books/NBK83105/ PMID 22855972
- [Derived] Kilicarslan N, Gurbuz H, Tasgoz FN, Karaca U, Karasu D, Gamli M. Factors influencing neonatal outcomes in twin pregnancies undergoing cesarean section: a cross-sectional study. Rev Assoc Med Bras (1992). 2023 May 19;69(5):e20221464. doi: 10.1590/1806-9282.20221464. eCollection 2023. PMID 37222324